CLINICAL TRIAL: NCT07057219
Title: StepuP: Steps Against the Burden of Parkinson's Disease
Brief Title: Steps Against the Burden of Parkinson's Disease
Acronym: StepuP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Neuroscience Research Australia (Other); VU University of Amsterdam (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Shake it up Australia Foundation (Unknown); Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Yoshiro Okubo, Conjoint Senior Lecturer, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: iRECS5114; 2022885 (Other Grant/Funding Number: The National Health and Medical Research Council)
Record Dates: First submitted 2025-05-19; First posted 2025-07-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease (PD)
Keywords: EEG; EMG; perturbation; VR; real-world gait; wearable device; gait; balance; falls
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speed-dependent treadmill training (SDTT) (Active Comparator): SDTT adjusts the treadmill's speed in real time to match an individual's walking pace, creating a dynamic and adaptive training environment. This approach simulates real-world walking conditions, promoting neuromuscular coordination, balance, and functional mobility. By tailoring speed to the user's natural gait, SDTT supports the development of efficient and more natural walking patterns. It has shown promise across clinical populations, including those with neurological disorders, musculoskeletal conditions, or recovering from injury. Its flexibility allows for progressive challenge as walking ability improves, making SDTT a valuable tool for optimising gait and mobility outcomes.
  Interventions: Other: Exercise
- SDTT+ perturbations + VR triggered adaptations (Experimental): The SDTT+ program combines speed-dependent treadmill training with perturbations and VR-triggered adaptations. Reactive gait responses are elicited through controlled accelerations and decelerations of treadmill belts, simulating real-life balance challenges.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — SDTT adjusts the treadmill's speed in real time to match an individual's walking pace, creating a dynamic and adaptive training environment. This approach simulates real-world walking conditions, promoting neuromuscular coordination, balance, and functional mobility. By tailoring speed to the user's natural gait, SDTT supports the development of efficient and more natural walking patterns. It has shown promise across clinical populations, including those with neurological disorders, musculoskeletal conditions, or recovering from injury. Its flexibility allows for progressive challenge as walking ability improves, making SDTT a valuable tool for optimising gait and mobility outcomes.
  Other Names: SDTT; Treadmill training; Gait training
  Arms: Speed-dependent treadmill training (SDTT)
Other: Exercise — The SDTT+ program combines speed-dependent treadmill training with perturbations and VR-triggered adaptations. Reactive gait responses are elicited through controlled accelerations and decelerations of treadmill belts, simulating real-life balance challenges.
  Other Names: SDTT+; VR; perturbation training; Treadmill training; Gait training
  Arms: SDTT+ perturbations + VR triggered adaptations

SUMMARY:
Parkinson's Disease Treadmill Training RCT Summary

Parkinson's disease (PD) affects over 10 million people globally. Despite optimal pharmacological treatment, approximately 70% of individuals experience unstable gait and falls, leading to loss of confidence, social isolation, fractures, and frequent hospitalisations. Treadmill training-especially when augmented by mechanical or virtual-reality perturbations-has shown promise in improving gait and reducing fall risk. However, the mechanisms underlying these benefits remain poorly understood, limiting the ability to personalise interventions effectively.

This randomised controlled trial (RCT) forms part of the broader Steps Against the Burden of Parkinson's Disease project (CT-IDs: 6ef2e427b002, 6ef2e427b003, 6ef2e427b004), comprising three harmonised but independently conducted RCTs. All sites follow a shared core protocol, allowing for pooled data analysis while preserving site-specific perturbation adaptations. Findings from this trial will be reported both independently and as part of the combined dataset.

In this trial, participants with PD will undergo 12 sessions of treadmill training, with or without virtual reality and perturbation-based adaptations. Assessments will be conducted at baseline, post-training, and follow-up. The intervention aims to enhance gait through improved sensorimotor integration and balance control. During the follow-up period, a smartphoneapp "Walking Tall" will be used to encourage continued exercises and long-term retention of training effects.

Biomechanical analyses will focus on changes in foot placement control. Neurophysiological outcomes will be examined using EEG and EMG, targeting reductions in beta-band EEG power and enhanced EEG-EMG coherence as markers of improved gait stability.

Recognising that laboratory-based improvements may not always translate to daily life, this study will also investigate gait self-efficacy as a potential moderator of transfer. Remote monitoring tools will capture real-world mobility outcomes over a week. Machine learning techniques will be employed to identify factors differentiating those who improve in both settings from those who do not. These insights will inform the development of personalised interventions capable of translating training effects into meaningful real-life outcomes.

DETAILED DESCRIPTION:
i. Rationale The rationale of this trial is that speed-dependent treadmill training (SDTT) improves gait in people with Parkinson's disease (PD) through enhanced sensorimotor integration, with cortical activity changes as underlying neural correlates. Additional benefits may be gained when treadmill training includes perturbations, which help train reactive balance responses. Furthermore, it is hypothesised that improvements in gait quality through SDTT can enhance gait self-efficacy, which may mediate or moderate the transfer of training effects to everyday mobility. Understanding these mechanisms is essential for personalising interventions and maximising real-world outcomes.

ii. Objectives

The objectives of the StepuP project are to:

1. Understand the kinematic and neural mechanisms that underlie improvements in gait due to treadmill training with and without mechanically and VR-triggered gait adaptations in people with PD.
2. Assess the extent to which gait improvements measured in the laboratory transfer to improvements in daily-life mobility.
3. Identify the mechanisms that support or limit the transfer of training effects from lab-based gait improvements to real-world mobility.
4. Determine for whom treadmill training improves gait characteristics in the lab and for whom it does not, and similarly, who benefits in terms of daily-life mobility.

Achieving these objectives will advance understanding of the variability in individual response to treadmill training, allowing more targeted and ultimately personalised interventions to improve outcomes in PD.

iii. Endpoints This trial will evaluate the effects of treadmill training with and without perturbations on gait performance and neural correlates in people with PD.

Primary endpoint:

> Change in gait speed under controlled treadmill conditions.

Secondary endpoints:

* Clinical outcomes: Changes in motor symptoms and function measured through clinical assessments.
* Kinematic outcomes: Changes in gait parameters such as step length and variability from baseline to follow-up.
* Neurophysiological outcomes: EEG and EMG markers, including changes in EEG beta power and EEG-EMG coherence.

Exploratory endpoints:

* Real-world gait metrics assessed via wearable sensors.
* Gait self-efficacy assessed with validated questionnaires to examine psychological influences on transfer.

These outcomes will help identify how and for whom treadmill training leads to meaningful, lasting improvements in mobility.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PD according to the MDS Criteria
2. Hoehn and Yahr stages I to III;
3. Movement Disorder Society-sponsored version of the Unified Parkinson Disease Rating Scale (MDS-UPDRS) gait sub-score of 1 or more
4. Signed informed consent to participation

Exclusion Criteria:

* Any known general health condition likely to interfere with or to pose a contraindication to non-medically supervised physical exercise.
* Moderate or severe depression (BDI-II ≥18)
* Cognitive impairment which may preclude the possibility to provide a fully informed consent to enrolment.
* Linguistic comprehension capacity less than 75% in ordinary conversation
* Severe psychiatric comorbidity which may interfere with compliance to the study protocol
* History of or current status of substance dependency
* Unable to walk less than 1 floor
* Thoracic pain in the last 4 weeks
* Currently enrolled in other interventional studies
* Implanted Deep Brain Stimulation device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Baseline (week 1), Post-Training (week 14), Follow-up (week 26)
  Comfortable walking speed overground

SECONDARY OUTCOMES:
Fall Events | Retrospective report at Baseline (week 1); ongoing reporting through Follow-up (week 26).
  The number of falls experienced and whether they resulted in injury will be recorded. This includes a 12-month retrospective report at baseline and ongoing reporting throughout the study.
EuroQol 5-Dimension (EQ-5D) Questionnaire | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  This quality-of-life instrument includes a descriptive profile and a visual analogue scale (VAS) to rate current health. The VAS ranges from 0 (the worst health imaginable) to 100 (the best health imaginable). Higher scores on the VAS indicate better health status.
Frailty Index (FI) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The Frailty Index assesses physical frailty based on five criteria: shrinking (unintentional weight loss), low physical endurance or energy (self-reported exhaustion), low physical activity, weakness (grip strength), and slow walking speed. Based on the number of criteria met (0 to 5), participants are classified into the following categories:
  Non-frail (0 criteria met) Pre-frail (1-2 criteria met) Frail (3 or more criteria met)
FACIT Fatigue Scale (Functional Assessment of Chronic Illness Therapy - Fatigue) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The FACIT Fatigue Scale measures self-reported fatigue and its impact on daily activities and functioning over the past week. Each item is scored on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Very much"). Total Score Range: 0 to 52. Higher scores indicate less fatigue and better functioning.
Visual Analogue Scale (VAS) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The VAS is used to assess subjective pain intensity or other symptom severity.
Foot placement kinematics | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  Three-dimensional motion capture will be used to evaluate gait and movement patterns, specicially the foot placement in relation to the centre of mass.
Timed Up and Go (TUG) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The TUG test assesses mobility, balance, and walking ability.
Two-Minute Walk Test (2MWT) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  This test measures functional exercise capacity by recording the distance walked in two minutes.
Mini-BESTest | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The Mini-BESTest evaluates dynamic balance across multiple domains of postural control.
Modified Gait Efficacy Scale (mGES) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The mGES measures confidence in walking under challenging everyday conditions.
Short Falls Efficacy Scale International (Short FES-I) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The Short Falls Efficacy Scale International is a 7-item questionnaire assessing concern about falling during a range of physical and social activities. Each item is scored from 1 (not at all concerned) to 4 (very concerned), resulting in a total score ranging from 7 to 28. Higher scores indicate greater concern about falling, which reflects a worse outcome.
Montreal Cognitive Assessment (MoCA) | Baseline (week 1), Follow-up (week 26).
  The MoCA evaluates cognitive function, including memory, attention, language, and executive functions. The MoCA consists of 30 points, with scores ranging from 0 to 30. Higher scores indicate better cognitive function, reflecting a better outcome.
Color Trail Test (CTT) | Baseline (week 1), Follow-up (week 26).
  The CTT assesses cognitive flexibility, visual attention, and processing speed. The CTT consists of two parts (CTT-1 and CTT-2), where participants are required to connect numbered circles in sequence, alternating between colours in the second part. Performance is measured by the time (in seconds) taken to complete each part. shorter completion times indicate better cognitive function, reflecting a better outcome.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS Part III) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The MDS-UPDRS Part III is the motor examination component of the Unified Parkinson's Disease Rating Scale developed by the Movement Disorder Society. It assesses motor signs of Parkinson's disease across 18 items (e.g., tremor, rigidity, bradykinesia, posture, gait), each rated on a 5-point scale from 0 (normal) to 4 (severe impairment).
  The total score ranges from 0 to 132. Higher scores indicate greater motor impairment, reflecting a worse outcome.
New Freezing of Gait Questionnaire (NFOGQ) | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The NFOGQ is a 9-item patient-reported instrument designed to assess the presence, severity, and impact of freezing of gait (FOG) in individuals with Parkinson's disease. Items are scored on a 5-point Likert scale ranging from 0 (absence or no impact) to 4 (severe or frequent impact).
  The total score ranges from 0 to 28, with higher scores reflecting more severe and frequent freezing episodes.
  Higher scores indicate worse freezing of gait symptoms, representing a worse outcome.
Daily Step Count | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The average number of steps taken per day will be recorded via wearable sensors.
Uninterrupted Walking Duration | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  Duration of uninterrupted walking bouts will be measured using wearable sensors.
Stride Time Variability | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  Stride-to-stride variability in walking rhythm will be derived from sensor data.
Gait Symmetry | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  The symmetry of gait parameters between left and right limbs will be calculated.
System Usability Scale (SUS) | Post-Training (week 14), Follow-up (week 26).
  Participants' acceptability and satisfaction with the intervention will be assessed via the SUS. The SUS is a 10-item questionnaire that assesses user satisfaction and perceived usability of a system or intervention. Each item is rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree).
  Raw item scores are converted to a composite score ranging from 0 to 100. Higher scores indicate better perceived usability and greater user satisfaction, reflecting a better outcome.
Physical Activity Enjoyment Scale (PACES) | Post-Training (week 14), Follow-up (week 26).
  Participants' acceptability and satisfaction with the intervention will be assessed via the PACES. The PACES is an 18-item questionnaire designed to assess enjoyment of physical activity. Each item is rated on a 7-point Likert scale (e.g., from "I enjoy it" to "I hate it"), with some items reverse-scored.
  The total score ranges from 18 to 126, with higher scores indicating greater enjoyment of physical activity, reflecting a better outcome.
Attitudes Towards Physical Activity | Post-Training (week 14), Follow-up (week 26).
  The Exercise Self-Efficacy Scale (ESES) will assess changes in attitudes toward physical activity. The ESES is a 10-item questionnaire that assesses confidence in engaging in physical activity despite common barriers. Each item is rated from 1 (not at all confident) to 4 (always confident).
  Total scores range from 10 to 40. Higher scores indicate greater confidence in the ability to exercise, reflecting a better outcome.
Participant experience | Post-Training (week 14), Follow-up (week 26).
  Semi-structured qualitative interviews will explore participant experiences, perceived barriers, enablers, and reasons for withdrawal. As this is a qualitative assessment, no numerical scale applies, and responses will be analysed using thematic analysis methods.
Beta band activity | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  EEG (electroencephalogram) will be used to measure brain activity by recording electrical signals from the scalp. It will assess beta band activity during walking to examine changes in cortical involvement associated with gait and training.
EEG-EMG coherency in the beta band | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  Coherency between EEG and EMG signals in the beta frequency band will be assessed during walking to evaluate changes in corticomuscular connectivity associated with gait and training.

OTHER OUTCOMES:
Fracture History | Baseline (week 1).
  The number and type of fractures sustained in the 12 months prior to baseline will be recorded.
Changes in medication | Baseline (week 1), Post-Training (week 14), Follow-up (week 26).
  All current medications (including antiparkinsonian and non-antiparkinsonian drugs) will be recorded at each study visit to monitor changes in use and assess potential side effects.
  Changes in medication will be categorised (e.g., dosage adjustments), and the number of participants with any change in medication will be reported.
Number of participants using mobility aids (indoors and outdoors) | Baseline (week 1), Follow-up (week 26).
  The use of mobility aids (e.g., cane, walker, rollator) will be documented separately for indoor and outdoor environments.
  The number and percentage of participants using walking aids will be reported at each time point.
Hand Grip Strength | Baseline (week 1).
  Grip strength will be assessed using a hand dynamometer as a proxy for overall strength and frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brodie, PhD, Study Chair — University of New South Wales; Yoshiro Okubo, PhD, Principal Investigator — Neuroscience Research Australia, University of New South Wales; Daniel Chan, PhD, MD, Principal Investigator — University of New South Wales; Luca Modenese, PhD, Principal Investigator — University of New South Wales; Frederic von Wegner, PhD, MD, Principal Investigator — University of New South Wales; Phu Hoang, PhD, MD, Principal Investigator — Neuroscience Research Australia; Husna Razee, PhD, Principal Investigator — University of New South Wales; Paulo Silva Pelicioni, PhD, Principal Investigator — University of New South Wales; Vicki Miller, Principal Investigator — Shake it up Australia Foundation; Carolyn Sue, PhD, MD, Principal Investigator — Neuroscience Research Australia; Martin Ostrowski, PhD, Principal Investigator — University of New South Wales; Mayna Ratanapongleka, Principal Investigator — Neuroscience Research Australia
Locations (1):
- Neuroscience Research Australia, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
The pseudonymized personal dataset corresponding to study participants who have opted in at the time of consent
Time Frame: The pseudonymized personal dataset corresponding to study participants who have opted in at the time of consent will be made available within two years of study completion
Access Criteria: Researchers comply with applicable data protection law, particularly Chapter V of the GDPR and the recommendations of the European Data Protection Board.
  Researchers submit an approved data management and intended use plan.
  Researchers approved by all sites including the University of New South Wales Human Research Ethics Committee.
URL: https://openneuro.org/